CLINICAL TRIAL: NCT03089047
Title: A Pilot Study on the Impact of Rejuvenated Autologous Blood Transfusion on VO2 Max in Healthy Subjects
Brief Title: Rejuvenated RBC and VO2 Max in Healthy Subjects
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Reagent shortage
Sponsor: Duke University (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Pro00078468
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-12

CONDITIONS: Erythrocyte Transfusion

STUDY DESIGN:
Intervention Model Description: Prospective randomized "healthy volunteer" study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Addition of rejuvesol will be performed by the blood bank and only they will know of group assignment
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rejuvenated RBC Transfusion (Experimental): Washed and Rejuvenated autologous blood
  Interventions: Biological: Transfusion of rejuvenated and washed autolgous RBCs
- Standard RBC Transfusion (Sham Comparator): Washed autologous blood (so as to maintain equivalent unit volume and Hct)
  Interventions: Biological: Transfusion of washed autolgous RBCs

INTERVENTIONS:
Biological: Transfusion of rejuvenated and washed autolgous RBCs — Rejuvenation refers to the process of adding a mix of solutes (Rejuvesol®, Citra Labs, Braintree, MA; consists of sodium pyruvate, inosine, adenine, mono- and dibasic sodium phosphate) to older, stored (i.e., 2-3 DPG-depleted) blood to immediately restore 2,3-DPG and ATP levels in the stored red blood cells15. Rejuvenation was originally developed to prolong the storage life of rare-phenotype RBC units. It is FDA-approved for use in RBC units stored in CPD, CPDA-1, and AS-1. The major contraindication for the use of Rejuvesol® is in RBC units stored for fewer than 6 days due to high baseline 2,3-DPG and ATP levels. Rejuvenated units must be washed prior to administration to remove residual Rejuvesol that is not approved for iv administration in such concentrations.
  Arms: Rejuvenated RBC Transfusion
Biological: Transfusion of washed autolgous RBCs — Autologous RBCs will be washed prior to transfusion to maintain blinding and equalize volume and Hct with the rejuvenated and washed intervention arm
  Arms: Standard RBC Transfusion

SUMMARY:
To compare the physiologic benefits of rejuvenated RBCs (rejRBCs) to standards RBCs (PRBCs), we will emulate critical conditions by safely maximizing stress on the cardiovascular system, in an elective, feasible volunteer study. Maximal oxygen uptake (VO2max) will be measured in an anemic, post-donation, pre-transfusion state, and also after transfusing 14-day-old, autologous blood randomized to standard storage or standard storage with rejuvenation. We hypothesize that transfusion of standard PRBCs is less effective at increasing oxygen delivery (measured by VO2max) compared with transfusion of rejRBCs.

DETAILED DESCRIPTION:
VISIT A ( - Screening) Written informed consent will be obtained from subjects who respond to an IRB-approved advertisement/flyer and fulfill eligibility requirements. The following video will help explain the study: vimeo.com/167291799. Individuals who respond to an IRB approved advertisement/flyer (uploaded to eIRB) will be given information about the study and asked to read an IRB approved consent form. An investigator or designee will obtain written informed consent from each individual participating in this study, after adequate explanation of the methods, objectives, and potential hazards of the study. The investigator or designee will also explain to the subjects that they are completely free to refuse to enter the study and free to withdraw from it at any time. A copy of the signed consent form will be given to the subject and will be shared with The Blood Connection to ensure proper labeling of autologous units.

After subjects have provided written informed consent, they will be asked to answer several questions in 2 written questionnaires (uploaded to eIRB) in order to confirm that they are eligible to donate blood. These questions are similar to those routinely asked to people prior to a blood donation. These are focused upon keeping the risks of blood donation to the lowest possible level. Subject will undergo screening lab tests for baseline hemoglobin, sickle cell trait, serum pregnancy tests only for women of child-bearing potential, ECG, exercise test. Subject will receive a phone confirmation from the investigator or delegated research staff after review of the screening lab results. Subject will bring a copy of the signed consent form to The Blood Connection if qualified.

VISIT B (Day 0 - Blood donation) The Blood Connection (TBC), Raleigh, NC, is registered and licensed by the US FDA and accredited by the American Association of Blood Banks (AABB) to manufacture RBCs and other blood products. Two units of blood will be withdrawn from each subject according to standards for double, AS-3, apheresis units, and will be marked for autologous donation, and purchased by Duke Transfusion Services, as arranged with the medical director of TBC (Robert Rainer, MD). RBC handling and storage will meet FDA and AABB standards; units will be stored with Duke Transfusion Services c/o Dr. Poisson.

VISIT C (Day 14 - "Anemic" VO2 max, Transfusion (Tx) and "post-Tx" VO2max)) Small amount of blood [3 lavender topped tubes] will be collected from subject to test for hemoglobin, type & screen and 1 cross match to verify the donated blood received from The Blood Connection belongs to the same subject who arrives at the appointed date at Duke facility

Anemic VO2max Three minutes of resting baseline measures will be recorded before the start of exercise. The subject will then begin to pedal the cycle ergometer at a cadence of 75 rpm. Resistance will be manually set according to a standardized, progressive protocol. A rating of perceived exertion (RPE) will be obtained at the end of each exercise stage. Vital signs will be recorded every 3 minutes, and ECG monitoring will be continuous. Exercise will be terminated when the subject reaches volitional fatigue. VO2max will be reported as the highest oxygen consumption averaged over two 30-second periods, which typically occurs in the last stage of the progressive maximal exercise test. Maximum heart rate will be the heart rate at or near VO2max. To minimize variability in VO2max testing procedures, the same 2 facilitators (an engineer/technician and a research staff) will be present at every test. Radial arterial access will be obtained for cardiac output monitoring (LiDCO pulse contour analysis) at this visit.

Tx and post-Tx VO2max Duke Transfusion Services will randomize each subject to receive 2 units of standard PRBCs or rejRBCs over 120 minutes using a standard infusion pump. All units will be washed to equalize the transfusion volumes; rejuvenation includes a mandatory washing step. Rejuvenation of donated blood will be done according to the procedures in the labeling of the Rejuvesol product. Vital signs will be monitored and recorded every 15 minutes. After a total 4-hour rest after completing the first VO2max testing, and a light snack, the exercise test will be repeated.

Laboratory testing: The p50 will be measured in one of the blood units transfused and in the subject before the exercise test. Radial arterial access will be obtained for serial cardiac output monitoring (LiDCO Pulse Contour Analysis, LiDCO Products, London, UK), arterial blood gas analysis and lactate measurement before and after transfusion, and after exercise testing. Final blood collected for a hemoglobin level will be done at the conclusion of blood transfusion. This is the final visit and participation is completed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Age 18-40 (the American College of Sports Medicine Guidelines for Exercise Testing defines this age group with no or no more than one coronary heart disease risk factor as low-risk for VO2 max testing)
* Habitual exerciser defined as ≥ 30 minutes of at least moderate or high intensity exercise ≥ 3 times per week. After consent, and at the subsequent screening visit, a VO2 max test will be performed, and subjects with a low value (< 35 mL/kg/min) will be excluded (screen failure). Based on our previous experience, we anticipate that up to 25% of the subjects will fall into this category; therefore, 10 subjects will be screened to obtain 6-8 participants who go on to donate their blood.
* Calculated total blood volume of at least 4,500 mL using an established formula:

  1. Men: (0.006012 x H3) + (14.6 x W) + 604 = TBV
  2. Women: (0.005835 x H3) + (15 x W) + 183 = TBV [H= Height in inches; W=Weight in pounds]
* Has access to transportation to visit the blood collection facility and to return to Duke for all study visits
* Weighs at least 130 pounds

Exclusion Criteria:

* Any significant acute or chronic medical illness or problem, including, but not limited to, diabetes, hypertension, cardiac disease, asthma, COPD
* Current or recent (last 60 days) tobacco or nicotine use
* History of sickle cell trait or disease or any other acquired or hereditary hematological abnormality
* History of fainting or other significant adverse reaction during phlebotomy or donation of blood
* Known prolonged QTc (or evidence of such at screening) defined as QTc >470 ms
* Known or suspected illicit drug or alcohol abuse
* Known or suspected HIV, Hepatitis B, or Hepatitis C infection
* History of thrombophilia or anticoagulant therapy
* Pregnancy
* Obesity defined as BMI>30
* Recent history of blood donation:

  1. Single whole blood unit donation within the past 8 weeks
  2. Double RBC donation by apheresis within the past 16 weeks
  3. Plasma donation by apheresis within the past 4 weeks
* Inadequate red blood cell mass evidenced by total blood volume <4500 mL (above) or screening hemoglobin <13.3 g/dL
* Known hypersensitivity to lithium compounds.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian J Welsby, BSc MBBS, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 subjects failed to meet baseline VO2max threshold, 1 had a below threshold hemoglobin prior to blood donation, and 1 enrolled in another study before completing baseline VO2max.
Period: Overall Study
Arm/Group | Rejuvenated RBC Transfusion | Standard RBC Transfusion
Started | 2 | 2
Completed | 1 | 2
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rejuvenated RBC Transfusion | Standard RBC Transfusion | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 2 | 3
VO2max [Mean (Standard Deviation); unit: ml/kg/min] | 44.80 (0) | 49.15 (9.97) | 47.70 (7.48)

OUTCOME MEASURES:

1. Primary Outcome: Change in VO2max
Description: Change in VO2max from "anemic" (pre-transfusion) VO2max and after transfusion of 2 units of either standard PRBCs or rej-PRBCs "post-Tx" VO2max.
Time Frame: Day 16 to Day 18 post transfusion
Population: Subjects who completed the study.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Rejuvenated RBC Transfusion | Standard RBC Transfusion
Number analyzed (Participants) | 1 | 2
ml/kg/min | 0.70 (0) | 6.05 (1.20)

2. Primary Outcome: Change in Lactate
Description: Change in lactate from "anemic" (pre-transfusion) VO2max and after transfusion of 2 units of either standard PRBCs or rej-PRBCs "post-Tx" VO2max
Time Frame: Day 16 to Day 18 post transfusion
Population: Data not collected.
Arm/Group | Rejuvenated RBC Transfusion | Standard RBC Transfusion
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in "Post-Tx" VO2max From Baseline
Description: Change in "post-Tx" (after transfusion) VO2max at day 18 from baseline.
Time Frame: Baseline to Day 18 post transfusion
Population: Subjects who completed the study.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Rejuvenated RBC Transfusion | Standard RBC Transfusion
Number analyzed (Participants) | 1 | 2
ml/kg/min | -1.90 (0) | -2.70 (2.40)

ADVERSE EVENTS:
Time Frame: 18 days
Arm/Group | Rejuvenated RBC Transfusion | Standard RBC Transfusion
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT03089047/Prot_SAP_000.pdf